CLINICAL TRIAL: NCT04051827
Title: A Phase 1, Open-Label, Multicenter, Drug-Drug Interaction Study of TAK-788 and Midazolam, a Sensitive CYP3A Substrate, in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Drug-Drug Interaction Study of TAK-788 and Midazolam in Participants With Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: TAK-788-1004; 2019-000725-44 (EudraCT Number); U1111-1225-0210 (Other: WHO)
Record Dates: First submitted 2019-08-05; First posted 2019-08-09 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Neoplasms
Keywords: Drug therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Midazolam; mobocertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Midazolam + TAK-788 (Experimental): Midazolam 3 mg, solution, orally, once on Days 1 and 24 and midazolam 1 mg, infusion, intravenously, once on Days 2 and 25 along with TAK-788 160 mg, capsule, orally, once daily from Day 3 through 30 in Cycle 1.
  Interventions: Drug: Midazolam; Drug: TAK-788
- Part B: TAK-788 (Experimental): TAK-788 160 mg, capsules, orally, once daily in a 28-day treatment cycle from Cycle 2 to Cycle 24, or until progressive disease (PD), intolerable toxicity, or another discontinuation criterion is met, whichever is sooner. Eligible participants from Part A may enter into Part B. Based on the investigator's opinion, if a participant continues to experience clinical benefit, treatment with TAK-788 may be continued after PD.
  Interventions: Drug: TAK-788

INTERVENTIONS:
Drug: Midazolam — Midazolam Oral Solution and Midazolam Intravenous Infusion.
  Arms: Part A: Midazolam + TAK-788
Drug: TAK-788 — TAK-788 Oral Capsules.
  Other Names: AP32788

SUMMARY:
The purpose of this study is to characterize the effect of repeated oral administration of TAK-788 160 milligram (mg) once daily on the single oral and intravenous dose pharmacokinetics (PK) of midazolam.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-788. The study will characterize the effect of repeated oral administration of TAK-788 160 mg on the single oral- and intravenous-dose PK of midazolam, and will assess the safety and tolerability of TAK-788 in participants with advanced NSCLC.

The study will enroll approximately 26 participants. The study will be conducted in 2 parts: Part A (Cycle 1: PK Cycle) and Part B (Cycle 2 to Cycle 24: Treatment Cycles). In Part A, participants will receive midazolam as an oral dose and intravenous infusion, along with oral dose of TAK-788 in a single 30-day cycle. After completion of Part A, eligible participants may enter Part B. In Part B, participants will continue to receive oral dose of TAK-788 that they were receiving and tolerating at the end of Part A in a 28-day treatment cycle for up to 23 cycles of treatment, or until progressive disease (PD), intolerable toxicity, or another discontinuation criterion is met. Based on the opinion of investigator, if a participant continue to experience clinical benefit, treatment with TAK-788 may be continued after PD.

This multi-center trial will be conducted in Australia, Singapore and the Netherlands. The overall time to participate in this study is 3 years. Participants will make multiple visits to the clinic and will be followed up for 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced NSCLC in which the participant is not a candidate for definitive therapy; or, the participant has recurrent or metastatic (Stage IV) disease.
2. Refractory or intolerant to standard available therapies.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
4. Minimum life expectancy of 3 months or more.
5. Adequate organ function as defined by the following criteria:

   * Total serum bilirubin less than or equal to (<=) 1.5*upper limit of normal (ULN) (<=3*ULN for participants with Gilbert syndrome or if liver function abnormalities are due to underlying malignancy)
   * Alanine aminotransferase and aspartate aminotransferase <=2.5*ULN (or <=5*ULN if liver function abnormalities are due to underlying malignancy)
   * Estimated creatinine clearance greater than or equal to (>=) 30 milliliter per minute (mL/min) (calculated by using the Cockcroft-Gault equation)
   * Serum albumin >= 2 gram/deciliter (g/dL)
   * Serum lipase/amylase <=1.5*ULN; and
   * Serum amylase <=1.5*ULN unless the increased serum amylase is due to salivary isoenzymes.
6. Adequate bone marrow function as defined by the following criteria:

   * Absolute neutrophil count >=1.5*10^9 per liter (/L)
   * Platelet count >=75*10^9/L; and
   * Hemoglobin >=9.0 g/dL.
7. Normal QT interval on screening electrocardiogram (ECG), defined as QT interval with Fridericia's correction (QTcF) of <= 450 millisecond (msec) in males or <= 470 msec in females. (as conducted and interpreted in accordance to local institutional practices and confirmed by principal investigator [PI]).
8. All toxicities from prior anticancer therapy must have resolved to <= Grade 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 or have resolved to baseline, at the time of first dose of TAK-788. Note: treatment-related Grade 2 or 3 alopecia and treatment-related Grade 2 peripheral neuropathy are allowed if deemed irreversible.
9. Suitable venous access for study-required blood sampling (that is, including for PK, pharmacodynamics, and clinical laboratory tests).

Exclusion Criteria:

1. Received a strong or moderate cytochrome P450 3A (CYP3A) inhibitor or strong or moderate CYP3A inducer within 2 weeks prior to the first dose of TAK-788.
2. Received small-molecule anticancer therapy (including but not limited to cytotoxic chemotherapy and investigational agents) within 2 weeks prior to the first dose of TAK-788.
3. Received antineoplastic monoclonal antibodies including check point inhibitors within 28 days of the first dose of TAK-788.
4. Received radiotherapy <=14 days prior to the first dose of TAK-788. However, participants are allowed to receive any of the following treatments up to 7 days prior to the first dose: (a) Stereotactic radiosurgery (SRS) (b) stereotactic body radiation therapy (SBRT) or (c) palliative radiation outside the chest and brain.
5. Major surgery within 28 days prior to the first dose of TAK-788. Minor surgical procedures, such as catheter placement or minimally invasive biopsy, are allowed.
6. Diagnosed with another primary malignancy other than NSCLC except for adequately treated non-melanoma skin cancer or cervical cancer in situ; definitively treated non-metastatic prostate cancer; or another primary malignancy and is definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.
7. Have known active brain metastases (have either previously untreated intracranial central nervous system (CNS) metastases or previously treated intracranial CNS metastases with radiologically documented new or progressing CNS lesions). Brain metastases are allowed if they have been treated with surgery and/or radiation and have been stable without requiring corticosteroids to control symptoms within 7 days before the first dose of TAK-788, and have no evidence of new or enlarging brain metastases.
8. Current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging) or leptomeningeal disease (symptomatic or asymptomatic).
9. Have uncontrolled hypertension. Participants with hypertension should be under treatment on study entry to control blood pressure.
10. Significant, uncontrolled, or active cardiovascular disease, including, but not limited to the following:

    * Myocardial infarction within 6 months prior to the first dose of study drug;
    * Unstable angina within 6 months prior to the first dose of study drug;
    * Congestive heart failure within 6 months prior to the first dose of study drug. Cardiac ejection fraction <50% by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA);
    * History of clinically significant (as determined by the treating physician) atrial arrhythmia;
    * Any history of ventricular arrhythmia; or
    * Cerebrovascular accident or transient ischemic attack within 6 months prior to the first dose of study drug.
11. Treatment with medications known to be associated with the development of torsades de pointes.
12. Gastrointestinal illness or disorder that could affect oral absorption of TAK-788 or midazolam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (8):
- Australia (4):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Peninsula and Southeast Oncology, Frankston, Victoria
  - Nucleus Network, Melbourne, Victoria
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam, North Holland
  - Universitair Medisch Centrum Groningen, Groningen
- Singapore (2):
  - The National University Cancer Institute - Singapore, Singapore
  - Raffles Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants.

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a346?idFilter=%5B%22TAK-788-1004%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in Australia, Singapore, and Netherlands from 23 December 2019 to 07 December 2021.
Pre-assignment Details: Participants with a historical diagnosis of locally advanced or metastatic non-small cell lung cancer (NSCLC) were enrolled in this 2-part study to receive midazolam oral solution along with mobocertinib (formerly TAK-788) capsule in Part A (Cycle 1) and mobocertinib capsule only in Part B (Cycle 2 to 19). After completion of Part A, eligible participants entered Part B to continue treatment with mobocertinib. As planned, combined safety data for Parts A and B was collected and reported.
Groups:
- Parts A and B: Midazolam + Mobocertinib: Midazolam 3 milligram (mg), solution, orally, once on Days 1 and 24 and midazolam 1 mg, infusion, intravenously, once on Days 2 and 25 along with mobocertinib 160 mg, capsule, orally, once daily from Day 3 through Day 30 in Cycle 1 (Month 1) in Part A. After completion of Part A, eligible participants continued treatment with mobocertinib in Part B to receive mobocertinib 160 mg, capsule, orally, once daily in a 28-day treatment cycle from Cycle 2 to Cycle 19 (Month 18).
Period: Overall Study
Arm/Group | Parts A and B: Midazolam + Mobocertinib
Started | 26
Completed | 0
Not Completed | 26
Not completed — Death | 1
Not completed — Withdrawal by Subject | 4
Not completed — Progressive disease | 16
Not completed — Physician Decision | 1
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all participants who received at least 1 dose of any study drug (mobocertinib or midazolam).
Groups:
- Parts A and B: Midazolam + Mobocertinib: Midazolam 3 mg, solution, orally, once on Days 1 and 24 and midazolam 1 mg, infusion, intravenously, once on Days 2 and 25 along with mobocertinib 160 mg, capsule, orally, once daily from Day 3 through Day 30 in Cycle 1 (Month 1) in Part A. After completion of Part A, eligible participants continued treatment with mobocertinib in Part B to receive mobocertinib 160 mg, capsule, orally, once daily in a 28-day treatment cycle from Cycle 2 to Cycle 19 (Month 18).
Arm/Group | Parts A and B: Midazolam + Mobocertinib
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (14.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 14
  Singapore | 7
  Netherlands | 5

OUTCOME MEASURES:

1. Primary Outcome: Part A, Cmax: Geometric Mean Maximum Observed Plasma Concentration (Cmax) for Midazolam Administered Orally With Mobocertinib (Cycle 1 Day 24) and Without Mobocertinib (Cycle 1 Day 1)
Description: As planned, this pharmacokinetic (PK) outcome measure was only assessed in Part A.
Time Frame: Cycle 1: Days 1 and 24 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length is equal to [=] 30 days)
Population: Pharmacokinetic (PK) evaluable population (Part A, Cycle 1) received protocol-specified dosing regimen without dose reductions prior to Day 26; had no dose interruptions within 1 week prior to Day 24; experienced no more than 1 day of dose interruption within first 14 days of mobocertinib; did not receive excluded concomitant medications through Day 26; and had sufficient midazolam concentration-time data to permit reliable estimation of PK parameters by noncompartmental analysis methods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part A: Midazolam Alone: Midazolam 3 mg, solution, orally, once on Day 1 in Cycle 1 (Month 1).
- Part A: Midazolam + Mobocertinib: Midazolam 3 mg, solution, orally, once on Day 24 along with mobocertinib 160 mg, capsule, orally, once daily from Day 3 through Day 30 in Cycle 1 (Month 1).
Arm/Group | Part A: Midazolam Alone | Part A: Midazolam + Mobocertinib
Number analyzed (Participants) | 13 | 13
nanogram per milliliter (ng/mL) | 17.0 (60.2) | 17.5 (60.7)
Statistical Analysis 1: Comparison: Part A: Midazolam Alone vs Part A: Midazolam + Mobocertinib; The ratios of geometric mean midazolam Cmax (in the presence vs absence of mobocertinib) and the associated 2-sided 90 percent (%) confidence intervals (CIs) were calculated on the basis of the within-patient variance using a mixed-effects analysis of variance (ANOVA) model fitting terms for treatment (midazolam in the absence and presence of mobocertinib); Test type: Other — Geometric Mean Ratio; Geometric Mean Ratio (GMR) = 1.03, 90% CI 2-sided [0.739 to 1.42] — The geometric mean ratio (GMR) of midazolam Cmax on Day 24 (with mobocertinib) versus on Day 1 (without mobocertinib) were calculated

2. Primary Outcome: Part A, AUC∞: Geometric Mean Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Midazolam Administered Orally With Mobocertinib (Cycle 1 Day 24) and Without Mobocertinib (Cycle 1 Day 1)
Description: As planned, this PK outcome measure was only assessed in Part A.
Time Frame: Cycle 1: Days 1 and 24 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length = 30 days)
Population: PK evaluable population. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Part A: Midazolam Alone | Part A: Midazolam + Mobocertinib
Number analyzed (Participants) | 13 | 12
nanogram*hour per milliliter (ng*h/mL) | 58.3 (61.0) | 39.0 (61.4)
Statistical Analysis 1: Comparison: Part A: Midazolam Alone vs Part A: Midazolam + Mobocertinib; The ratios of geometric mean midazolam AUC∞ (in the presence vs absence of mobocertinib) and the associated 2-sided 90% CIs were calculated on the basis of the within-patient variance using a mixed-effects ANOVA model fitting terms for treatment (midazolam in the absence and presence of mobocertinib); Test type: Other — Geometric Mean Ratio; Geometric Mean Ratio (GMR) = 0.676, 90% CI 2-sided [0.532 to 0.859] — The GMR of midazolam AUC∞ on Day 24 (with mobocertinib) versus on Day 1 (without mobocertinib) were calculated

3. Primary Outcome: Part A, Cmax: Geometric Mean Maximum Observed Plasma Concentration (Cmax) for Midazolam Administered Intravenously With Mobocertinib (Cycle 1 Day 25) and Without Mobocertinib (Cycle 1 Day 2)
Description: As planned, this PK outcome measure was only assessed in Part A.
Time Frame: Cycle 1: Days 2 and 25 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length = 30 days)
Population: PK evaluable population (Part A, Cycle 1) received protocol-specified dosing regimen without dose reductions prior to Day 26; had no dose interruptions within 1 week prior to Day 24; experienced no more than 1 day of dose interruption within first 14 days of mobocertinib; did not receive excluded concomitant medications through Day 26; and had sufficient midazolam concentration-time data to permit reliable estimation of PK parameters by noncompartmental analysis methods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part A: Midazolam Alone: Midazolam 1 mg, infusion, intravenously, once on Day 2 in Cycle 1 (Month 1).
- Part A: Midazolam + Mobocertinib: Midazolam 1 mg, infusion, intravenously, once on Day 25 along with mobocertinib 160 mg, capsule, orally, once daily from Day 3 through Day 30 in Cycle 1 (Month 1).
Arm/Group | Part A: Midazolam Alone | Part A: Midazolam + Mobocertinib
Number analyzed (Participants) | 13 | 13
ng/mL | 70.8 (151.0) | 92.2 (132.0)
Statistical Analysis 1: Comparison: Part A: Midazolam Alone vs Part A: Midazolam + Mobocertinib; The ratios of geometric mean midazolam Cmax (in the presence vs absence of mobocertinib) and the associated 2-sided 90% CIs were calculated on the basis of the within-patient variance using a mixed-effects ANOVA model fitting terms for treatment (midazolam in the absence and presence of mobocertinib); Test type: Other — Geometric Mean Ratio; Geometric Mean Ratio (GMR) = 1.30, 90% CI 2-sided [0.886 to 1.92] — The GMR of midazolam Cmax on Day 25 (with mobocertinib) versus on Day 2 (without mobocertinib) were calculated

4. Primary Outcome: Part A, AUC∞: Geometric Mean Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Midazolam Administered Intravenously With Mobocertinib (Cycle 1 Day 25) and Without Mobocertinib (Cycle 1 Day 2)
Description: As planned, this PK outcome measure was only assessed in Part A.
Time Frame: Cycle 1: Days 2 and 25 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length = 30 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: Midazolam Alone | Part A: Midazolam + Mobocertinib
Number analyzed (Participants) | 13 | 12
ng*h/mL | 90.4 (113.0) | 71.6 (96.0)
Statistical Analysis 1: Comparison: Part A: Midazolam Alone vs Part A: Midazolam + Mobocertinib; [analysis description as in outcome 2, analysis 1]; Test type: Other — Geometric Mean Ratio; Geometric Mean Ratio (GMR) = 0.837, 90% CI 2-sided [0.673 to 1.04] — The GMR of midazolam AUC∞ on Day 25 (with mobocertinib) versus on Day 2 (without mobocertinib) were calculated

5. Primary Outcome: Part A, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Midazolam Administered Orally With Mobocertinib (Cycle 1 Day 24) and Without Mobocertinib (Cycle 1 Day 1)
Description: As planned, this PK outcome measure was only assessed in Part A for midazolam 3 mg oral solution.
Time Frame: Cycle 1: Days 1 and 24 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length = 30 days)
Population: PK evaluable population (Part A, Cycle 1) received protocol-specified dosing regimen without dose reductions prior to Day 26; had no dose interruptions within 1 week prior to Day 24; experienced no more than 1 day of dose interruption within first 14 days of mobocertinib; did not receive excluded concomitant medications till completion of PK sampling (Day 26); and had sufficient midazolam concentration-time data to permit reliable estimation of PK parameters by noncompartmental analysis methods.
Measure: Median (Full Range); unit: hour
Arm/Group | Part A: Midazolam Alone | Part A: Midazolam + Mobocertinib
Number analyzed (Participants) | 13 | 13
hour | 0.517 [0.467 to 2.00] | 0.533 [0.250 to 1.00]

6. Primary Outcome: Part A, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Midazolam Administered Intravenously With Mobocertinib (Cycle 1 Day 25) and Without Mobocertinib (Cycle 1 Day 2)
Description: As planned, this PK outcome measure was only assessed in Part A for midazolam 1 mg intravenous infusion.
Time Frame: Cycle 1: Days 2 and 25 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length = 30 days)
Population: as for outcome 5
Measure: Median (Full Range); unit: hour
Arm/Group | Part A: Midazolam Alone | Part A: Midazolam + Mobocertinib
Number analyzed (Participants) | 13 | 13
hour | 0.0500 [0.00 to 1.00] | 0.0500 [0.00 to 0.500]

7. Secondary Outcome: Part A and B: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Part A:From Day 1 up to 30 days after the last dose of study drug in Cycle 1 (up to 2 months);Part B:From Day 1 of Cycle 2 up to 30 days after the last dose of study drug in Cycle 19 (up to Month 19) (Cycle length, Part A= 30 days; Part B=28 days)
Population: The safety population was defined as all participants who received at least 1 dose of any study drug (mobocertinib or midazolam). Since treatment with mobocertinib was intended to continue without any modification from Part A into Part B, therefore it was planned to analyze the combined safety data (Parts A and B).
Measure: Count of Participants; unit: Participants
Groups:
- Parts A and B: Midazolam + Mobocertinib: Midazolam 3 mg, solution, orally, once on Days 1 and 24 and midazolam 1 mg, infusion, intravenously, once on Days 2 and 25 along with mobocertinib 160 mg, capsule, orally, once daily from Day 3 through Day 30 in Cycle 1 in Part A. After completion of Part A, eligible participants continued treatment with mobocertinib in Part B to receive mobocertinib 160 mg, capsule, orally, once daily in a 28-day treatment cycle from Cycle 2 to Cycle 19 (Month 18).
Arm/Group | Parts A and B: Midazolam + Mobocertinib
Number analyzed (Participants) | 26
Participants | 26

8. Secondary Outcome: Part A and B: Number of Participants With Clinically Significant Change From Baseline in Laboratory Values
Description: The clinically significant change from baseline in laboratory values was assessed by the investigator.
Time Frame: Part A: Day 1 of Cycle 1; Part B: Day 1 of every Cycle (Cycle 2 to Cycle 19) (Cycle length, Part A=30 days; Part B =28 days)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Parts A and B: Midazolam + Mobocertinib
Number analyzed (Participants) | 26
Participants
  Blood creatinine increased | 7
  Amylase increased | 3
  Lipase increased | 3

9. Secondary Outcome: Part A and B: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Time Frame: Part A: Day 1 up to Day 26 in Cycle 1; Part B: Day 1 of every Cycle (Cycle 2 to Cycle 19) (Cycle length, Part A=30 days; Part B =28 days)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Parts A and B: Midazolam + Mobocertinib
Number analyzed (Participants) | 26
Participants | 0

ADVERSE EVENTS:
Time Frame: TEAEs were adverse events that started from Day 1 up to 30 days after the last dose of study drug in Cycle 1 (up to 2 months) for Part A and from Day 1 of Cycle 2 up to 30 days after the last dose of study drug in Cycle 19 (up to Month 19) for Part B (Cycle length, Part A= 30 days and Part B=28 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Since treatment with mobocertinib was intended to continue without any modification from Part A into Part B, therefore it was planned to analyze the combined safety data (Parts A and B).
Arm/Group | Parts A and B: Midazolam + Mobocertinib
All-Cause Mortality (participants affected / at risk) | 4/26
Serious Adverse Events (participants affected / at risk) | 20/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Parts A and B: Midazolam + Mobocertinib (N=26)
Arrhythmia (Cardiac disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nausea (Gastrointestinal disorders) | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pneumonia (Infections and infestations) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Spinal cord compression (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Parts A and B: Midazolam + Mobocertinib (N=26)
Abdominal pain (Gastrointestinal disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4
Amylase increased (Investigations) | 3
Anaemia (Blood and lymphatic system disorders) | 5
Angular cheilitis (Gastrointestinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Blood creatinine increased (Investigations) | 7
Chills (General disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Decreased appetite (Metabolism and nutrition disorders) | 13
Dehydration (Metabolism and nutrition disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 25
Dizziness (Nervous system disorders) | 4
Dry mouth (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 6
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Fatigue (General disorders) | 13
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Headache (Nervous system disorders) | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Insomnia (Psychiatric disorders) | 2
Lethargy (Nervous system disorders) | 2
Lipase increased (Investigations) | 3
Mouth ulceration (Gastrointestinal disorders) | 2
Mucosal inflammation (General disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Paronychia (Infections and infestations) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4
Pyrexia (General disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 9
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Stomatitis (Gastrointestinal disorders) | 4
Taste disorder (Nervous system disorders) | 2
Urinary tract infection (Infections and infestations) | 4
Vomiting (Gastrointestinal disorders) | 9
Weight decreased (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT04051827/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT04051827/SAP_001.pdf